CLINICAL TRIAL: NCT03918044
Title: Elective and Non-elective Cesarean Section and the Risk for Obesity Among Young Male Conscripts: a Population-based Cohort and Matched-sibling Analysis.
Brief Title: Obesity Among Young Adult Males Born With Cesarean Section.
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Daniel Berglind, Principal Investigator, Karolinska Institutet
Other Study IDs: 20190405
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2019-08

CONDITIONS: Caesarean Section; Obesity; Cesarean Section Complications
Keywords: Obesity; Cesarean Section; Vaginal Delivery; Elective Cesarean Section; Non-elective Cesarean Section
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous research has suggested that cesarean section may be associated with an increased risk of developing obesity in childhood, adolescence and adulthood. Yet, previous studies have been small or unable to differentiate between elective and non-elective cesarean section. Therefore, using a population-based cohort the purpose is to examine the associations between vaginal delivery, elective and non-elective cesarean section on the risk of developing obesity in young adulthood among Swedish young singleton males. Using the Swedish medical birth registry, the recorded mode of delivery and indication of delivery which will be matched to those males who perform military conscription, where their body mass index is recorded. The investigators hypothesize that there will be an elevated risk of obesity in those born with non-elective cesarean section, as a function of confounding, while those born with elective cesarean section will not have a higher risk of obesity than those born with vaginal delivery.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth.
* Retrievable from medical birth registry.

Exclusion Criteria:

* No available information on mode of delivery.
* Not conscripted.
* Extreme values at conscription.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All singleton born in Sweden between 1982 and 1987.
Sampling Method: Probability Sample
Enrollment: 97291 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Categories of body mass index | Measured at conscription (~18 years of age)
  World health organisation categories of body mass index: underweight BMI<18.5, normal weight BMI 18.5-24.9, overweight BMI 25-29.9 and obese BMI>30. Weight at conscription was measured using standardized scales and height was assessed using stadiometers in a standardized manner.

SECONDARY OUTCOMES:
Continuous body mass index | Measured at conscription (~18 years of age)
  Measured continuous body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Ahlqvist VH, Persson M, Magnusson C, Berglind D. Elective and nonelective cesarean section and obesity among young adult male offspring: A Swedish population-based cohort study. PLoS Med. 2019 Dec 6;16(12):e1002996. doi: 10.1371/journal.pmed.1002996. eCollection 2019 Dec. PMID 31809506

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/44/NCT03918044/Prot_SAP_002.pdf